CLINICAL TRIAL: NCT03029442
Title: The Efficacy of Denosumab to Prevent Bone Loss in Ambulatory and Non-ambulatory Motor-Incomplete Patients With Subacute Spinal Cord Injury
Brief Title: The Efficacy of Denosumab in Incomplete Patients Spinal Cord Injury
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study ended early due to COVID-19
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Kessler Institute for Rehabilitation (Industry)
Responsible Party: Principal Investigator, William A. Bauman, M.D., Director, Clinical Investigator, National Center of Excellence for the Medical Consequences of Spinal Cord Injury, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BAU-16-057
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Secondary Osteoporosis; Spinal Cord Injury
Keywords: Spinal Cord Injury; Denosumab; Osteoporosis; Dual Energy X-ray Absorptiometry
MeSH Terms: conditions — Spinal Cord Injuries; Osteoporosis | interventions — Denosumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Denosumab, AIS Grade C (non-ambulatory) (Experimental): 8 subjects with AIS grade C will be randomized to receive Denosumab (Prolia 120mg SC) administered at baseline and 6 months.
  Interventions: Drug: Denosumab (Prolia)
- Placebo, AIS Grade C (non-ambulatory) (Placebo Comparator): 8 subjects with AIS grade C will be randomized to the placebo group and will receive the identical volume of normal saline at parallel time points.
  Interventions: Other: Placebo (normal saline)
- Denosumab, AIS Grade D (ambulatory) (Experimental): 8 subjects with AIS grade D will be randomized to receive Denosumab (Prolia 120mg SC) administered at baseline and 6 months.
  Interventions: Drug: Denosumab (Prolia)
- Placebo, AIS Grade D (ambulatory) (Placebo Comparator): 8 subjects with AIS grade D will be randomized to the placebo group and will receive the identical volume of normal saline at parallel time points.
  Interventions: Other: Placebo (normal saline)

INTERVENTIONS:
Drug: Denosumab (Prolia) — In clinical trials, denosumab (Amgen Inc., Thousand Oaks, CA), has been shown to be more potent in reducing osteoclastosis and function than bisphosphonates. The dose of denosumab chosen for our protocol in patients after acute SCI will be the same dose that has been shown to be efficacious to treat postmenopausal osteoporosis (60 mg SQ q 6 months).
  Other Names: Xgeva
  Arms: Denosumab, AIS Grade C (non-ambulatory); Denosumab, AIS Grade D (ambulatory)
Other: Placebo (normal saline) — Identical Denosumab volume of normal saline
  Arms: Placebo, AIS Grade C (non-ambulatory); Placebo, AIS Grade D (ambulatory)

SUMMARY:
The purpose of this study is to determine the usefulness of a drug, denosumab, to prevent the loss of bone in participants legs due to SCI. This drug is FDA approved to treat osteoporosis in women after menopause who have an increased risk for fractures, to treat women receiving certain treatments for breast cancer who have an increased risk of fractures, and to treat bone loss in men receiving certain treatments for prostate cancer who have increased risk for fractures. This drug is considered experimental for the purpose of this study. Study participation will last for approximately 12 months (6 study visits total), visits will range from1-4.5 hours depending on the number of tests that need to be completed. The study is a double-blinded placebo trail in which the participant will be randomly assigned to on of two groups, Denosumab injections or placebo - inactive salt solution injections.

DETAILED DESCRIPTION:
The primary objective of this study is to test the efficacy of a potent anti-resorptive agent, denosumab [receptor activator of nuclear factor-κB ligand (RANKL) antibody; Amgen Inc.] to preserve bone mass at the hip and knee and trabecular connectivity at the knee after subacute motor-incomplete SCI [American Spinal Injury Association (AIS) neurological classification scale C and D] at the James J. Peters VA Medical Center (JJPVAMC) and Kessler Institute for Rehabilitation (KIR). A randomized, double-blind, placebo-controlled, parallel group trial will be performed in thirty-two subjects with acute, motor-incomplete SCI (≤6 months) who have been admitted to JJPVAMC or the KIR. Denosumab (60 mg SC) will be administered at baseline, 6, and 12 months; the placebo group will receive normal saline subcutaneously. Denosumab will be administered as soon as possible, but up to 24 weeks, after SCI. The last dose of denosumab and placebo will be administered at 6 months, with the anticipated effect of the drug to persist and inhibit bone resorption at least until the 12 month time point.

ELIGIBILITY:
Inclusion Criteria:

1. Motor incomplete SCI [American Spinal Injury Association Impairment Scale (AIS) grades C and D];
2. Duration of injury < 6-months; and
3. Males between the ages of 18 and 65 years old and females between the ages of 18 and 50 years old.

Exclusion Criteria:

1. Extensive life-threatening injuries in addition to SCI;
2. Acute fracture or extensive bone trauma;
3. History of prior bone disease (Paget's hyperparathyroidism, osteoporosis, etc.)
4. Post-menopausal women;
5. Men with known hypogonadism prior to SCI;
6. Anabolic or Steroid hormonal therapy; within the past year and longer than six months;
7. Hyperthyroidism;
8. Cushing's disease or syndrome;
9. Severe underlying chronic disease;
10. History of chronic alcohol abuse;
11. Diagnosis of Hypocalcemia;
12. Pregnancy;
13. Existing dental condition/dental infection;
14. Diagnosis of heterotopic ossification at the hip and/or knee region and receiving a bisphosphonates [e.g. alendronate sodium (Fosamax) or etidronate disodium (Didronel)] that will no longer make participants eligible to receive the study medication/placebo but are still eligible to complete follow-up outcome measures as described in the work schedule;
15. Current diagnosis of cancer or history of cancer; and
16. Any patient receiving moderate or high dose corticosteroids (>40 mg/d prednisone or an equivalent dose of other corticosteroid) for longer than one week, not including drug administered in an attempt to preserve neurological function at the time of acute SCI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
areal bone mineral density (aBMD) by dual energy X-ray absorptiometry (DXA) | Prior to denosumab or placebo administration and 18 months after denosumab or placebo administration
  Efficacy of denosumab to prevent aBMD loss at the distal femur and proximal tibia

SECONDARY OUTCOMES:
volumetric BMD (vBMD) and microarchitecture by peripheral quantitative computed tomography | Prior to denosumab or placebo administration and 12 months after denosumab or placebo administration
  Efficacy of denosumab to prevent vBMD loss and microarchitecture deterioration at the distal femur and proximal tibia

CONTACTS AND LOCATIONS:
Overall Officials: William A Bauman, M.D., Principal Investigator — James J. Peters VA Medical Center; Steven C Kirshblum, M.D., Principal Investigator — Kessler Institute for Rehabilitation
Locations (2):
- United States (2):
  - Kessler Institute for Rehabilitation, West Orange, New Jersey
  - James J. Peters VA Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No
An IPD is not desired by the investigators and is not part of the regulatory guidelines at the participating institutions

REFERENCES:
- [Background] Gifre L, Vidal J, Carrasco JL, Muxi A, Portell E, Monegal A, Guanabens N, Peris P. Denosumab increases sublesional bone mass in osteoporotic individuals with recent spinal cord injury. Osteoporos Int. 2016 Jan;27(1):405-10. doi: 10.1007/s00198-015-3333-5. Epub 2015 Sep 30. PMID 26423406